CLINICAL TRIAL: NCT05027919
Title: Assessing a Clinically-meaningful Opioid Withdrawal Phenotype
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00279895; 1R01DA052937 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Opioid Withdrawal; Opioid Use Disorder; Opioid Craving
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Hydromorphone; Naloxone; lofexidine

STUDY DESIGN:
Masking Description: The order of medication pre-treatment during the two Naloxone Challenges will be blinded to participants and the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Within-subject design (Other): All participants will undergo the same study design, which includes hydromorphone stabilization (days 1-5), two naloxone challenges (scheduled during morphine stabilization), lofexidine-assisted taper (days 6-10), and transition to aftercare (day 11).
  Interventions: Drug: Hydromorphone; Drug: Naloxone + lofexidine pretreatment; Drug: Naloxone + placebo pretreatment; Drug: Lofexidine

INTERVENTIONS:
Drug: Hydromorphone — Up to 120mg oral per day in q4 dosing to manage withdrawal
Drug: Naloxone + lofexidine pretreatment — 0.2-0.4mg naloxone injection during the Naloxone challenge + pretreatment with oral lofexidine (25% of max daily dose scheduled during lofexidine taper)
Drug: Naloxone + placebo pretreatment — 0.2-0.4mg naloxone injection during the Naloxone challenge
Drug: Lofexidine — Oral Lofexidine dosed per FDA label (4 times daily) on days 6 through 10.

SUMMARY:
Evaluate individual differences in the expression of opioid withdrawal symptoms in persons with opioid use disorder (OUD) while completing a clinically-indicated medication taper.

DETAILED DESCRIPTION:
Individuals who have opioid use disorder and are interested in being tapered off of opioids will be admitted to a residential research unit for an 11-day period. All participants will be maintained on morphine for 5 days. During this period participants will complete 2 sessions (on two different days) wherein participants will receive an intramuscular injection of naloxone to precipitate a short withdrawal syndrome. Participants will take a capsule prior to both sessions that will contain either placebo or the opioid withdrawal medication lofexidine. Beginning on day 6 participants will be tapered off of morphine using lofexidine (as clinically indicated). At the end of the study all participants will be able to transition to buprenorphine maintenance or receive oral naltrexone and an injection of Vivitrol (extended release naltrexone), consistent with standard of care practices. Investigators will collect a variety of biological samples and questionnaire ratings during the study and primary outcomes will be measures of withdrawal collected throughout the study. Investigators will use these data to learn more about why individuals express opioid withdrawal symptoms differently, which will help inform how to change current treatment practices to be more effective for persons with OUD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years - 65 year old
* Opioid-positive urine sample
* Current opioid use disorder with evidence of physical dependence
* Interest in undergoing opioid taper

Exclusion Criteria:

* Evidence of physical dependence on alcohol or benzodiazepines that requires medical intervention
* Being pregnant or breastfeeding
* Enrolled in methadone or buprenorphine maintenance treatment
* Clinically significant hypotension (<90/60mmHg) or bradycardia (<45bpm)
* History of myocardial infarction
* Subjects who are positive for hepatitis B surface antigen and/or hepatitis C antibody with liver function tests outside the normal range (persons with a positive hepatitis C antibody and normal liver functions tests are NOT excluded from the study)
* Significant mental health or physical disorder, or life circumstances, that is expected to interfere with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Withdrawal severity during lofexidine taper | Days 6 through 10
  Withdrawal severity as assessed by the Subjective Opioid Withdrawal Scale. (The score range is 0 through 64) with higher score indicating more severe withdrawal.
Withdrawal severity during naloxone challenge | Days 1 through 5
  Withdrawal severity as assessed by the Subjective Opioid Withdrawal scale scores (The range is 0 through 64) with higher score indicating more severe withdrawal. Collected during two naloxone challenges (pretreatment with lofexidine and pretreatment with placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dunn, Ph.D, M.B.A., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No